CLINICAL TRIAL: NCT06760949
Title: A Single Center Prospective Controlled Study of Direct Anterior Approach and Posterior Lateral Approach in the Treatment of Femoral Neck Fractures in Elderly Patients
Brief Title: Comparative Study on Surgical Approaches for Elderly Femoral Neck Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Provincial Hospital (Other)
Collaborators: Fujian Provincial Hospital Emergency Center (Unknown)
Responsible Party: Principal Investigator, CHEN JIAN, Principal investigator, Fujian Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fujian Trauma Center
Record Dates: First submitted 2024-12-20; First posted 2025-01-07 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Function; Pain
Keywords: femoral neck fractures; direct anterior approach; hemiarthroplasty
MeSH Terms: conditions — Pain; Femoral Neck Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DAA group (Experimental): Patients with femoral neck fractures undergoing DAA-HA.
  Interventions: Procedure: Direct anterior approach hemiarthroplasty
- PLA group (Active Comparator): Patients with femoral neck fractures undergoing PLA-HA.
  Interventions: Procedure: Posterior lateral approach hemiarthroplasty

INTERVENTIONS:
Procedure: Direct anterior approach hemiarthroplasty — Direct anterior approach hemiarthroplasty
  Arms: DAA group
Procedure: Posterior lateral approach hemiarthroplasty — Posterior lateral approach hemiarthroplasty
  Arms: PLA group

SUMMARY:
A prospective controlled study was conducted to include patients who received hip replacement surgery for femoral neck fractures at the National Regional Trauma Center in Fujian Province from February 2023 to August 2024. Patients were randomly divided into the DAA group and the PLA group based on different surgical methods for a 3-month follow-up to compare the outcomes of the two groups. The main observation results include Harris hip joint function score (preoperative, postoperative 1 week, 1 month, 3 months), VAS pain score (preoperative, postoperative 1 week, 1 month, 3 months), and secondary observation results include surgical time, intraoperative blood loss, blood transfusion rate, difference in HB before and after surgery, difference in CK before and after surgery, perioperative complications, difference in length of both lower limbs after surgery, postoperative drainage volume, postoperative ICU occupancy rate, ICU length of stay, and total length of stay.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 80 years old;
2. Diagnosed with unilateral femoral neck fracture through imaging examination;
3. Patients who can tolerate surgery and agree to undergo surgery;
4. Undergoing hemiarthroplasty (HA) for the first time;
5. Able to walk independently and have intact cognitive function before the injury.

Exclusion Criteria:

1. Bilateral femoral neck fractures;
2. Patients with pathological fractures;
3. Hip dysplasia, rheumatoid osteoarthritis, or other hip disorders;
4. Patients with systemic or localized infections or inflammatory reactions at the surgical site;
5. Patients with other lower limb fractures or severe injuries to other parts of the body; Patients with a history of previous hip surgery.

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 102 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Harris hip joint function score | 1 week, 1 month, and 3 months after surgery
  Scores range from 100 to 0, with 90-100 being excellent, 80-89 being good, 70-79 being acceptable, and ≤69 being poor.
VAS pain score | 1 week, 1 month, and 3 months after surgery
  The highest score is 10 and the lowest score is 0, with the following interpretations: 0 points indicating no pain; 1-3 points indicating mild pain with little impact on daily life; 4-6 points indicating moderate pain affecting daily life and sleep; 7-9 points indicating severe pain significantly affecting quality of life; and 10 points indicating unbearable, extreme pain.

SECONDARY OUTCOMES:
Operative time | Intraoperative
Intraoperative bleeding volume | Intraoperative
Intraoperative blood transfusion rate | Intraoperative
Hemoglobin value | Preoperative and postoperative 1 day
Blood creatine kinase value | Preoperative and postoperative 1 day
Incidence of complications | Perioperative period
Difference in length of both lower limbs | 3 days after surgery
Postoperative drainage volume | 24 hours after surgery
Hospital stay | The duration (in days) from admission to discharge, estimated to be no more than 21 days at most.
Mortality | 3 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Provincial Hospital Trauma Center, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No
Because of unit regulations.

REFERENCES:
- [Result] Dahm F, Aichmair A, Dominkus M, Hofstaetter JG. Incidence of lateral femoral cutaneous nerve lesions after direct anterior approach primary total hip arthroplasty - a literature review. Orthop Traumatol Surg Res. 2021 Dec;107(8):102956. doi: 10.1016/j.otsr.2021.102956. Epub 2021 May 4. PMID 33962046
- [Result] Zhao G, Zhu R, Jiang S, Xu N, Bao H, Wang Y. Using the anterior capsule of the hip joint to protect the tensor fascia lata muscle during direct anterior total hip arthroplasty: a randomized prospective trial. BMC Musculoskelet Disord. 2020 Jan 11;21(1):21. doi: 10.1186/s12891-019-3035-9. PMID 31926554
- [Result] Ugland TO, Haugeberg G, Svenningsen S, Ugland SH, Berg OH, Pripp AH, Nordsletten L. Biomarkers of muscle damage increased in anterolateral compared to direct lateral approach to the hip in hemiarthroplasty: no correlation with clinical outcome : Short-term analysis of secondary outcomes from a randomized clinical trial in patients with a displaced femoral neck fracture. Osteoporos Int. 2018 Aug;29(8):1853-1860. doi: 10.1007/s00198-018-4557-y. Epub 2018 May 22. PMID 29789919
- [Result] Dimitriou D, Helmy N, Hasler J, Flury A, Finsterwald M, Antoniadis A. The Role of Total Hip Arthroplasty Through the Direct Anterior Approach in Femoral Neck Fracture and Factors Affecting the Outcome. J Arthroplasty. 2019 Jan;34(1):82-87. doi: 10.1016/j.arth.2018.08.037. Epub 2018 Sep 3. PMID 30262445
- [Result] Oba T, Inaba Y, Saito I, Fujisawa T, Saito T. Risk factors for prolonged operative time in femoral neck fracture patients undergoing hemiarthroplasty through direct anterior approach. J Orthop Sci. 2018 Nov;23(6):977-981. doi: 10.1016/j.jos.2018.07.003. Epub 2018 Aug 4. PMID 30087014
- [Result] Trinh TQ, Ferrel JR, Pulley BR, Fowler TT. Short-term Outcomes of Femoral Neck Fractures Treated With Hemiarthroplasty Using the Anterior Approach. Orthopedics. 2015 Dec;38(12):e1091-7. doi: 10.3928/01477447-20151120-05. PMID 26652329
- [Result] Ding ZC, Zeng WN, Rong X, Liang ZM, Zhou ZK. Do patients with diabetes have an increased risk of impaired fracture healing? A systematic review and meta-analysis. ANZ J Surg. 2020 Jul;90(7-8):1259-1264. doi: 10.1111/ans.15878. Epub 2020 Apr 7. PMID 32255244
- [Result] Jiao H, Xiao E, Graves DT. Diabetes and Its Effect on Bone and Fracture Healing. Curr Osteoporos Rep. 2015 Oct;13(5):327-35. doi: 10.1007/s11914-015-0286-8. PMID 26254939
- [Result] Jia P, Bao L, Chen H, Yuan J, Liu W, Feng F, Li J, Tang H. Risk of low-energy fracture in type 2 diabetes patients: a meta-analysis of observational studies. Osteoporos Int. 2017 Nov;28(11):3113-3121. doi: 10.1007/s00198-017-4183-0. Epub 2017 Aug 9. PMID 28795239
- [Result] Saxer F, Studer P, Jakob M, Suhm N, Rosenthal R, Dell-Kuster S, Vach W, Bless N. Minimally invasive anterior muscle-sparing versus a transgluteal approach for hemiarthroplasty in femoral neck fractures-a prospective randomised controlled trial including 190 elderly patients. BMC Geriatr. 2018 Sep 21;18(1):222. doi: 10.1186/s12877-018-0898-9. PMID 30241509
- [Result] Verzellotti S, Candrian C, Molina M, Filardo G, Alberio R, Grassi FA. Direct anterior versus posterolateral approach for bipolar hip hemiarthroplasty in femoral neck fractures: a prospective randomised study. Hip Int. 2020 Nov;30(6):810-817. doi: 10.1177/1120700019872117. Epub 2019 Aug 26. PMID 31450987
- [Result] Renken F, Renken S, Paech A, Wenzl M, Unger A, Schulz AP. Early functional results after hemiarthroplasty for femoral neck fracture: a randomized comparison between a minimal invasive and a conventional approach. BMC Musculoskelet Disord. 2012 Aug 8;13:141. doi: 10.1186/1471-2474-13-141. PMID 22873207
- [Result] Carlson VR, Ong AC, Orozco FR, Lutz RW, Duque AF, Post ZD. The Direct Anterior Approach Does Not Increase Return to Function Following Hemiarthroplasty for Femoral Neck Fracture. Orthopedics. 2017 Nov 1;40(6):e1055-e1061. doi: 10.3928/01477447-20170925-08. Epub 2017 Oct 3. PMID 28968478
- [Result] Chung YY, Lee SM, Baek SN, Park TG. Direct Anterior Approach for Total Hip Arthroplasty in the Elderly with Femoral Neck Fractures: Comparison with Conventional Posterolateral Approach. Clin Orthop Surg. 2022 Mar;14(1):35-40. doi: 10.4055/cios21008. Epub 2022 Jan 21. PMID 35251539
- [Result] Bucs G, Dande A, Patczai B, Sebestyen A, Almasi R, Not LG, Wiegand N. Bipolar hemiarthroplasty for the treatment of femoral neck fractures with minimally invasive anterior approach in elderly. Injury. 2021 Mar;52 Suppl 1:S37-S43. doi: 10.1016/j.injury.2020.02.053. Epub 2020 Feb 21. PMID 32115214
- [Result] Kunkel ST, Sabatino MJ, Kang R, Jevsevar DS, Moschetti WE. A systematic review and meta-analysis of the direct anterior approach for hemiarthroplasty for femoral neck fracture. Eur J Orthop Surg Traumatol. 2018 Feb;28(2):217-232. doi: 10.1007/s00590-017-2033-6. Epub 2017 Aug 29. PMID 28852880
- [Result] van der Sijp MPL, van Delft D, Krijnen P, Niggebrugge AHP, Schipper IB. Surgical Approaches and Hemiarthroplasty Outcomes for Femoral Neck Fractures: A Meta-Analysis. J Arthroplasty. 2018 May;33(5):1617-1627.e9. doi: 10.1016/j.arth.2017.12.029. Epub 2017 Dec 29. PMID 29398259
- [Result] Florschutz AV, Langford JR, Haidukewych GJ, Koval KJ. Femoral neck fractures: current management. J Orthop Trauma. 2015 Mar;29(3):121-9. doi: 10.1097/BOT.0000000000000291. PMID 25635363
- [Result] Leonardsson O, Rolfson O, Rogmark C. The surgical approach for hemiarthroplasty does not influence patient-reported outcome : a national survey of 2118 patients with one-year follow-up. Bone Joint J. 2016 Apr;98-B(4):542-7. doi: 10.1302/0301-620X.98B4.36626. PMID 27037438
- [Result] Berggren M, Stenvall M, Englund U, Olofsson B, Gustafson Y. Co-morbidities, complications and causes of death among people with femoral neck fracture - a three-year follow-up study. BMC Geriatr. 2016 Jun 3;16:120. doi: 10.1186/s12877-016-0291-5. PMID 27260196
- [Result] Neyisci C, Erdem Y, Bilekli AB, Bek D. Direct Anterior Approach Versus Posterolateral Approach for Hemiarthroplasty in the Treatment of Displaced Femoral Neck Fractures in Geriatric Patients. Med Sci Monit. 2020 Jan 21;26:e919993. doi: 10.12659/MSM.919993. PMID 31961830
- [Result] Spina M, Luppi V, Chiappi J, Bagnis F, Balsano M. Direct anterior approach versus direct lateral approach in total hip arthroplasty and bipolar hemiarthroplasty for femoral neck fractures: a retrospective comparative study. Aging Clin Exp Res. 2021 Jun;33(6):1635-1644. doi: 10.1007/s40520-020-01696-9. Epub 2020 Sep 10. PMID 32910422
- [Result] Huang XT, Liu DG, Jia B, Xu YX. Comparisons between Direct Anterior Approach and Lateral Approach for Primary Total Hip Arthroplasty in Postoperative Orthopaedic Complications: A Systematic Review and Meta-Analysis. Orthop Surg. 2021 Aug;13(6):1707-1720. doi: 10.1111/os.13101. Epub 2021 Aug 5. PMID 34351056
- [Result] JUDET J, JUDET R. The use of an artificial femoral head for arthroplasty of the hip joint. J Bone Joint Surg Br. 1950 May;32-B(2):166-73. doi: 10.1302/0301-620X.32B2.166. No abstract available. PMID 15422013
- [Result] Langlois J, Delambre J, Klouche S, Faivre B, Hardy P. Direct anterior Hueter approach is a safe and effective approach to perform a bipolar hemiarthroplasty for femoral neck fracture: outcome in 82 patients. Acta Orthop. 2015 Jun;86(3):358-62. doi: 10.3109/17453674.2014.1002987. Epub 2015 Jan 13. PMID 25583401
- [Result] Kannan A, Kancherla R, McMahon S, Hawdon G, Soral A, Malhotra R. Arthroplasty options in femoral-neck fracture: answers from the national registries. Int Orthop. 2012 Jan;36(1):1-8. doi: 10.1007/s00264-011-1354-z. Epub 2011 Sep 20. PMID 21931966
- [Result] Antapur P, Mahomed N, Gandhi R. Fractures in the elderly: when is hip replacement a necessity? Clin Interv Aging. 2011;6:1-7. doi: 10.2147/CIA.S10204. Epub 2010 Dec 20. PMID 21472086
- [Result] Sterling RS. Gender and race/ethnicity differences in hip fracture incidence, morbidity, mortality, and function. Clin Orthop Relat Res. 2011 Jul;469(7):1913-8. doi: 10.1007/s11999-010-1736-3. PMID 21161737

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT06760949/Prot_SAP_000.pdf
  • Informed Consent Form (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT06760949/ICF_001.pdf